CLINICAL TRIAL: NCT02830191
Title: Therapeutic Drug Monitoring (TDM) of Cyclosporine in Kidney Transplant Patients by Dried Blood Spot Assay. Interest and Feasibility.
Acronym: CICLOSPOT
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 14-050
Record Dates: First submitted 2016-07-06; First posted 2016-07-12 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2016-07

CONDITIONS: Kidney Transplantation
Keywords: Cyclosporine, Dried blood spot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Ciclosporin A (CsA) is an immunosuppressive drug used in organs and tissues transplantations (kidney, heart, liver, bone marrow ...) to prevent rejection, and in different autoimmune or inflammatory diseases. A therapeutic drug monitoring (TDM) is required during a CsA treatment. It is justified by a narrow therapeutic range between efficiency and nephrotoxicity, and by large intra- and interindividual pharmacokinetic variability. TDM of CsA is conventionally performed by determining residual concentration, and sometimes concentration at 2 hours after administration. TDM of CsA is currently performed by venous sampling on ethylenediaminetetraacetic acid (EDTA). Dried blood spot (DBS) sampling could be a particularly interesting alternative to conventional blood sampling. With DBS, capillary blood is obtained from a finger prick by the patient himself, and the blood drop obtained is deposited on filter paper, which can be stored at room temperature and then be sent to the laboratory by mail.

This sampling method has several advantages : it requires small blood volumes, it is less invasive than conventional venous sampling, sampling can be performed by the patient himself at home few days before the consultation, and the results of the analysis can be available to the clinician on the day of consultation, allowing dose adjustment more quickly.

Several studies have been published in recent years using DBS sampling method, for various drugs such as antimalarials, antiepileptics, antiretrovirals, metformin, benzodiazepines, or immunosuppressants. Only one clinical validation study of TDM of CsA using DBS method was published by Wilhelm et al. (2013) in a population of 38 patients who received allogeneic stem cell transplant recipients. The results showed excellent correlation between the concentrations determined by the two sampling methods.

The investigators propose an observational study at the University Hospital of Caen for clinical validation of DBS sampling for TDM of CsA in kidney transplantation, for which there are no data published. During a nephrology consultation, for each patient, venous and finger prick blood samples are simultaneously collected. CsA assays were performed by liquid chromatography-tandem mass spectrometry (LC-MS/MS) for the two sampling methods. A specific LC-MS/MS assay method applied for DBS samples was developed and validated for this study (DBS/LC-MS/MS). Correlation between the results obtained from the two sampling methods will be evaluated, on at least 100 samples. Patients have to answer a questionnaire to assess pain and comfort of DBS sampling, and feasibility of self-sampling at home by this method. The aim of this clinical validation study of DBS sampling is the establishment of the systematic TDM of CsA for renal transplant patients by DBS sampling at the University Hospital of Caen.

ELIGIBILITY:
Inclusion Criteria:

* Adult Patient (18 years or older) treated with CsA and monitored for dose adjustment
* Kidney transplantation
* Not objecting to participate in study

Exclusion Criteria:

* Objecting to the additional sample by finger prick
* Anticoagulant treatment
* Hemostatic disorder (risk of hematoma)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Renal transplant patients treated with cyclosporine at nephrology department of the University Hospital of Caen.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2014-11; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Correlation between CsA concentrations determined from DBS sampling and conventional venous sampling for each patient (coefficient correlation, Bland-Altman difference plot) | 8 months

SECONDARY OUTCOMES:
Comparison of pain, comfort and practicality of the two sampling methods by a patient questionnaire. | 8 months

IPD SHARING:
Plan to Share IPD: Yes